CLINICAL TRIAL: NCT01523028
Title: Influence of Breakfast Consumption on Chlorogenic Acid Metabolism in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11.12.NRC
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Coffee, bread and honey (Experimental): 200 mL coffee + 2 bread rolls + honey
  Interventions: Other: Soluble Coffee
- Coffee, bread and peanut butter (Experimental): 200 mL coffee + 1 bread roll + peanut butter
  Interventions: Other: Soluble Coffee
- 200 mL black coffee (Experimental)
  Interventions: Other: Soluble Coffee

INTERVENTIONS:
Other: Soluble Coffee — Amounts of chlorogenic acids will be normalized to body weight (3.1 mg CA / kg BW). Coffee will be reconstituted in 200 mL hot water and consumed 3 times in a row (min 1-week interval), alone or with a breakfast:
  * 200 mL coffee or
  * 200 mL coffee + 2 bread rolls + honey
  * 200 mL coffee + 1 bread roll + peanut butter

SUMMARY:
Data and knowledge gathered on bioavailability of coffee phenolics is becoming more and more important, hence underlying the importance of better understanding the fate of these potential health promoting antioxidants. However, some analytical barriers as well as some key aspects of metabolism still remain to be fully elucidated to get the full picture of coffee metabolism and bioavailability. One aspect addressed in the present study is the impact of food matrix in modulating absorption, plasma appearance and urinary excretion of coffee bioactives.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Aged 20-44 years
* Caucasian origin
* Body mass index (BMI) 19-25 kg/m2
* Used to drinking coffee (similar to study coffee) on a daily basis
* Being able to tolerate a 48-hour coffee abstinence
* Normal oral glucose tolerance test
* Having signed the informed consent form

Exclusion Criteria:

* Taking medication or dietary supplements
* Smoking
* Performing a competitive sport
* Having metabolic disorders
* Long gut transit time (>24 h)
* Blood donor
* Irregularity in menstrual cycle (for women)
* Pregnancy (for women)
* Subject who cannot be expected to comply with the study procedures.
* Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sum of plasma areas under the curve of coffee phenolics | Measurements over 24h after coffee ingestion

SECONDARY OUTCOMES:
Plasma AUC, Cmax and Tmax of individually measured coffee chlorogenic and phenolic acids | Measurements done over 24h after coffee ingestion
Urinary excretion of coffee chlorogenic and phenolic acids expressed as % ingested dose | Measurements done over 24h after coffee ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kaiserslautern, Kaiserslautern, Germany